CLINICAL TRIAL: NCT02992535
Title: Effect of Intense Pulse Light (IPL) Treatment on Tear Film Osmolarity in Dry Eye Disease (DED) With Meibomian Gland Dysfunction (MGD).
Brief Title: Effect of Intense Pulse Light (IPL) Treatment on Tear Film Osmolarity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carones Ophthalmology Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLEUROPE1
Record Dates: First submitted 2016-12-02; First posted 2016-12-14 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Intense pulse light therapy (E-Schwin)
  Interventions: Device: Intense Pulse Light Energy delivery (IPL)

INTERVENTIONS:
Device: Intense Pulse Light Energy delivery (IPL)

SUMMARY:
Evaluate changes in tear film osmolarity and other DED signs/symptoms following treatment with IPL.

DETAILED DESCRIPTION:
Prospective study design among subjects with MGD and qualifying for IPL therapy.

Study testing done at baseline visit when subjects are scheduled for IPL therapy. Measurements will be made on day 15 (prior to second IPL sitting), Day 45 (prior to third IPL setting), Day 75 (fourth IPL setting) and Day 105 as needed (30 days after IPL setting 4).

Subjects willing to come for follow up visits as scheduled and may not have instilled any artificial tears 2 hours prior to study measurements.

No history of ocular infection or corneal degeneration/dystrophy No history of corneal refractive surgery and/or change in ocular medications in the last 2 months

ELIGIBILITY:
Inclusion Criteria:

* Dry eye
* MGD

Exclusion Criteria:

* No history of ocular infection or corneal degeneration/dystrophy
* No history of corneal refractive surgery
* No change in ocular medications in the last 2 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tear film osmolarity change | Measurements will be made on day 15 (prior to second IPL sitting), Day 45 (prior to third IPL setting), Day 75 (fourth IPL setting) and Day 105 as needed (30 days after IPL setting 4).

IPD SHARING:
Plan to Share IPD: Undecided